CLINICAL TRIAL: NCT06197009
Title: A Randomized, Double-blinded, Phase II, Placebo-controlled Study to Evaluate the Safety and Efficacy of SCT650C in Participants With Axial Spondyloarthritis
Brief Title: Efficacy and Safety of SCT650C in Participants With Axial Spondyloarthritis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCT650C-MRCT-2-02
Record Dates: First submitted 2023-12-11; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Axial Spondyloarthritis
MeSH Terms: conditions — Axial Spondyloarthritis

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo Group /Group1 (Placebo Comparator): Induction: Placebo s.c. every 2 weeks. Maintenance: 160mg SCT650C s.c. every 4 weeks
  Interventions: Drug: SCT650C
- SCT650C low dose Group /Group 2 (Active Comparator): Induction: 160mg SCT650C s.c. every 2 weeks. Maintenance: 160mg SCT650C s.c. every 4 weeks
  Interventions: Drug: SCT650C
- SCT650C medium dose Group /Group3 (Active Comparator): Induction: 320mg SCT650C s.c. every 2 weeks. Maintenance: 320mg SCT650C s.c. every 4 weeks
  Interventions: Drug: SCT650C
- SCT650C high dose Group /Group 4 (Active Comparator): Induction: 320mg SCT650C s.c. every 2 weeks. Maintenance: 160mg SCT650C s.c. every 4 weeks
  Interventions: Drug: SCT650C

INTERVENTIONS:
Drug: SCT650C — Administered SC
  Other Names: Recombinant anti-IL-17A antibody

SUMMARY:
The purpose of this study is to assess efficacy, safety, pharmacokinetics and immunogenicity of subcutaneous SCT650C in patients with Axial Spondyloarthritis

DETAILED DESCRIPTION:
This is a multicenter, Phase II, double-blinded, placebo-controlled study to evaluate the safety and efficacy of SCT650C in Participants with Axial Spondyloarthritis. This study includes 4 periods (Screening period, Loading period, Maintenance period and Follow-up period), and 168 participants in 4 groups (Group 1, 2, 3 and 4).

ELIGIBILITY:
Inclusion Criteria:

1. An Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written Informed Consent form is signed and dated by the participant.
2. Participant is considered reliable and capable of adhering to the protocol (e.g., able to understand and complete diaries), visit schedule, and medication intake according to the judgment of the Investigator.
3. Participant is male or female and at least 18 years of age.
4. Participant has a documented diagnosis of adult-onset AS as defined by documented radiologic evidence (X-ray) fulfilling the Modified New York criteria for AS (1984) of at least 3 months' symptom duration and age of onset <45 years.
5. Participant has moderate to severe active disease at the Screening Visit as defined by each of the following:

   1. BASDAI score ≥4
   2. Spinal pain score ≥4 on a 0 to 10 numeric rating scale (NRS) (from BASDAI Item 2)
6. Participants must have at least 1 of the following:

   1. inadequate response to NSAID therapy
   2. intolerance to administration of at least 1 NSAID
   3. contraindication(s) to NSAID therapy An inadequate response to NSAID is defined as not improving after 4 weeks of using NSAID therapy at the recommended dose or failing to respond to at least 2 NSAIDs at the recommended dose for 2 weeks each.
7. Participants who are regularly taking NSAIDs/COX-2 inhibitors as part of their SPA therapy are required to be on a stable dose for at least 14 days before Baseline and should remain on a stable dose up to week 16.
8. Participants taking corticosteroids must be on an average daily dose of ≤10mg/day prednisone or equivalent for at least 14 days before Baseline and should remain on a stable dose up to week 16.
9. Participants taking Methotrexate (MTX, ≤25mg/week), sulfasalazine (up to 3g/day) or hydroxychloroquine (up to 400mg per day total) are allowed to continue their medication if the dose has been stable dose for at least 4 weeks before randomization. Dose, dosing schedule, and route of administration (oral or subcutaneous) should remain stable up to week 16.
10. Subject may have prior treatment TNF inhibitor (TNFi), which must have used no more than 2 TNFi and must have been discontinued.
11. Female participants must be postmenopausal (at least 1 year; to be confirmed hormonally as part of the screening process, if less than 2 years since last menstrual period), permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy) or, if of childbearing potential (and engaged in sexual activity that could result in procreation), must be willing to use a highly effective method of contraception up to 40 weeks after the last administration of IMP, and have a negative pregnancy test at Visit 1 (Screening) and immediately prior to the first dose. The following methods are considered highly effective when used consistently and correctly.

    1. progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
    2. combined (estrogen and progestogen) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal)
    3. intrauterine device (IUD)
    4. intrauterine hormone-releasing system (IUS)
    5. bilateral tubal occlusion
    6. vasectomized partner (where postvasectomy testing had demonstrated sperm clearance)
    7. Sexual abstinence if it is in accordance with a participant's preferred and common lifestyle.

Participants who use abstinence as a form of birth control must agree to abstain from heterosexual intercourse until 40 weeks after the final dose of IMP. Study personnel must confirm the continued use of abstinence is still in accordance with the participant's lifestyle at regular intervals during the study.

Male participants with a partner of childbearing potential must be willing to use a condom when sexually active, until 40 weeks after the last administration of IMP.

Exclusion Criteria:

1. Female participant who is breastfeeding, pregnant, or planning to become pregnant during the study or within 40 weeks following the final dose of IMP. Male participant planning a partner pregnancy during the study or within 40 weeks following the final dose.
2. Participant has participated in another study of a medication under investigation within the last 3 months or at least 5 half-lives of the IMP, whichever is greater, or is currently participating in another study of a medication under investigation. Participants who participated in any clinical trial but were enrolled in placebo group and did not receive any IMP in the prior study are eligible for this study.
3. Participant has received any IL-17 response modifier.
4. Participant has received more than 3 bDMARDs to treat axSpA.
5. Participant has a known hypersensitivity to any excipients of SCT650C.
6. Participant has total ankylosis of the spine or a diagnosis of any other inflammatory arthritis e.g., RA, systemic lupus erythematosus, sarcoidosis, psoriatic arthritis, or reactive arthritis. Participants with a diagnosis of Crohn's disease or ulcerative colitis are allowed if they have no active symptomatic disease at Screening or Baseline.
7. Participant has a secondary noninflammatory condition (e.g., osteoarthritis, fibromyalgia) that in the Investigator's opinion is symptomatic enough to interfere with the evaluation of the effect of study drug on the participant's primary diagnosis of active SpA.
8. Participant has:

   1. A history of chronic or recurrent infections (e.g., more than 3 episodes requiring systemic antibiotics or antivirals during the preceding year). Minor illnesses like common cold or transient, localized infections that may have been treated with a short course of antibiotic therapy (up to 7 days) need not be counted in this assessment.
   2. A serious or life-threatening infection within the 6 months prior to the Baseline Visit (including herpes zoster) or hospitalization for any infection in the last 6 months.
   3. Any current sign or symptom that may indicate an active infection (except for common cold) or has had an infection requiring systemic antibiotics within 2 weeks prior to Baseline.
   4. A high risk of infection in the Investigator's opinion (e.g., participants with leg ulcers, indwelling urinary catheter, prior prosthetic joint infection at any time, participants who are permanently bedridden or wheelchair assisted).
9. Participant has a history of or current clinically active infection with Histoplasma, Coccidiodes, Paracoccidioides, Pneumocystis, nontuberculous mycobacteria (NTMB), Blastomyces, or Aspergillus or current active Candidiasis (local or systemic)
10. Participant has acute or chronic viral hepatitis B or C or human immunodeficiency virus (HIV) infection. Participants who have evidence of, or test positive for, hepatitis B or hepatitis C are excluded as follows:

    1. A positive test for the hepatitis B virus (HBV) is defined as: 1) positive for hepatitis B surface antigen (HBsAg+), or 2) HBsAg is negative, HBcAb is positive and HBV-DNA test results ≥ the upper limit of the reference value of each center or need antiviral treatment.
    2. A positive test for the hepatitis C virus (HCV) is defined as: 1) positive for hepatitis C antibody (anti-HCV Ab), and 2) positive via a confirmatory test for HCV (for example, HCV polymerase chain reaction).
11. Participants with known TB infection, at high risk of acquiring TB infection, with latent TB infection (LTBI), or current or history of NTMB infection.
12. Participant has a primary immunosuppressive condition, including taking immunosuppressive therapy following an organ transplant or has had a splenectomy.
13. Participants with concurrent malignancy or a history of malignancy (including surgically resected uterine/cervical carcinoma-in-situ) during the past 5 years will be excluded with the following exceptions that may be included:

    1. One squamous cell carcinoma of the skin (stage T1 maximum) successfully excised or ablated only (other treatments, i.e., chemotherapy, do not apply) with no signs of recurrence or metastases for more than 2 years prior to Screening.
    2. ≤3 excised or ablated basal cell carcinomas of the skin.
    3. Actinic keratosis(-es).
    4. Squamous cell carcinoma-in-situ of the skin successfully excised or ablated more than 6 months prior to the Screening.
14. Participant has a history of a lymphoproliferative disorder including lymphoma or current signs and symptoms suggestive of lymphoproliferative disease.
15. Participant has a history of demyelinating disease (including myelitis) or neurologic symptoms suggestive of demyelinating disease.
16. Participant has a current or recent history, as determined by the Investigator, of severe, progressive, and/or uncontrolled renal, hepatic hematological, endocrine, pulmonary, cardiac (e.g., congestive heart failure New York Heart Association [NYHA] Grade 3 and 4), gastrointestinal (GI) (note: participants with active peptic ulcer disease are excluded; participants with a history of peptic ulcer disease are allowed), or neurological disease.
17. Participants have a history of uncompensated heart failure, fluid overload, or myocardial infarction, or evidence of new-onset ischemic heart disease or in the opinion of the Investigator other serious cardiac disease, within 12 weeks prior to Baseline.
18. Participant has >2x upper limit of normal (ULN) of any of the following: alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), or >ULN total bilirubin (≥1.5xULN total bilirubin if known Gilbert's syndrome). If participant has elevations only in total bilirubin that is>ULN and <1.5xULN, fractionate bilirubin to identify possible undiagnosed Gilbert's syndrome (i.e., direct bilirubin <35%).

    An isolated elevation between 2xULN and <3xULN of ALP is acceptable in the absence of an identified exclusionary medical condition.

    Tests that result in ALT, AST, or ALP up to 25% above the exclusion limit may be repeated for confirmation during the Screening Period. Upon retesting, participants whose ALT, AST, or ALP remain above the thresholds defined above, should not be randomized.

    For randomized participants with a Baseline result >ULN for ALT, AST, ALP, or total bilirubin, a Baseline diagnosis and/or the cause of any clinically meaningful elevation must be understood and recorded in the electronic Case Report form (eCRF).

    If a participant has >ULN ALT, AST, or ALP that does not meet the exclusion limit at Screening, repeat the tests, if possible, prior to dosing to ensure there is no further ongoing clinically relevant increase. In case of a clinically relevant increase, inclusion of the participant must be discussed with the Medical Monitor.
19. Participants with clinically significant laboratory abnormalities (e.g., creatinine >1.5xULN, neutropenia <1.5x109/L, hemoglobin <8.5g/dL, lymphocytes <1.0 x109/L, white blood cell (WBC) count <3.0x109, platelets <100 x109/L). Individual screening tests for which the results are in error, borderline, or indeterminate for inclusion in the study, can be repeated once for confirmation during the Screening Period if they are within 25% of the exclusion limit. Upon retesting, participants whose results remain outside this threshold should not be randomized.
20. Participant has an estimated glomerular filtration rate (GFR) as measured by Chronic Kidney Disease Epidemiology Collaboration <60mL/min/1.73m2 [GFR (male)=(140-age)ⅹWeight/serum creatinineⅹ1.23; GFR (female)=(140-age)ⅹWeight/serum creatinineⅹ1.04].
21. Participant has a 12-lead ECG with changes considered to be clinically significant upon medical review (e.g., QT corrected for heart rate [QTc] using Fridericia's correction [QTcF] >450ms, bundle branch block, evidence of myocardial ischemia).
22. Participant has received any live (includes attenuated) vaccination within the 8 weeks prior to Baseline (12 months prior to Baseline for the TB Bacille Calmette-Guérin [BCG] vaccine) (e.g., inactivated influenza and pneumococcal vaccines are allowed but nasal influenza vaccination is not permitted). Live vaccines are not allowed during the study or for 40 weeks after the final dose of IMP.

    Live vaccines include, but are not limited to the following:
    1. Anthrax vaccine
    2. Intranasal influenza vaccine
    3. Measles-mumps-rubella (MMR) vaccine
    4. Polio live oral vaccine (OPV)
    5. Smallpox vaccine
    6. Tuberculosis BCG vaccine (within 12 months prior to Baseline)
    7. Typhoid live oral vaccine
    8. Varicella vaccine
    9. Yellow fever vaccine
23. Participant has any other condition which, in the Investigator's judgment, would make the participant unsuitable for inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Axial Spondyloarthritis Reporting Adverse Events (AEs), Serious Adverse Events (SAEs), and Treatment Emergent Adverse Events (TEAEs) | 48 Weeks
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
  A serious adverse event (SAE) is any untoward medical occurrence that at any dose:
  Results in death Is life-threatening Requires in patient hospitalisation or prolongation of existing hospitalisation Is a congenital anomaly or birth defect Is an infection that requires treatment parenteral antibiotics Other important medical events which based on medical or scientific judgement may jeopardise the patients, or may require medical or surgical intervention to prevent any of the above.
Percentage of Participants Achieving an Assessment of Spondyloarthritis International Society 40 (ASAS40) Response | week 16
  The ASAS40 response was defined as relative improvements of at least 40% and absolute improvement of at least 2 units on a 0 to 10 Numeric Rating Scale (NRS), where 0 is "not active" and 10 is "very active" in at least 3 of the 4 domains: Patient's Global Assessment of Disease Activity (PGADA), Pain assessment (total spinal pain NRS score), Function (Bath Ankylosing Spondylitis Functional Index (BASFI)), Inflammation (mean of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) questions 5 and 6 concerning morning stiffness intensity and duration) and no worsening at all in the remaining domain.
  Note: Participants with missing data or who discontinue study treatment prior to Week 12 were counted as non-responders.

SECONDARY OUTCOMES:
Percentage of Participants With Axial Spondyloarthritis International Society 20% Response Criteria (ASAS20) at Week 16 | week 16
  The ASAS20 response was defined as an improvement of at least 20% and absolute improvement of at least 1 unit on a 0 to 10 NRS, where 0 is "not active" and 10 is "very active" in at least 3 of the 4 domains: PGADA, Pain assessment (total spinal pain NRS scores), Function (BASFI), Inflammation (mean of BASDAI questions 5 and 6 concerning morning stiffness intensity and duration) and absence of deterioration in the potential remaining domain [deterioration was defined as a relative worsening of at least 20% and an absolute worsening of at least 1 unit].
  Note: Participants with missing data or who discontinue study treatment prior to Week 12 were counted as non-responders.
Change From Baseline in Ankylosing Spondylitis Disease Activity Score - C-Reactive Protein (ASDAS [CRP]) at Week 16 | week 16
  The ASDAS was calculated as the sum of the following components:
  0.121 x Back pain (BASDAI question 2 result) 0.058 x Duration of morning stiffness (BASDAI question 6 result) 0.110 x PGADA 0.073 x Peripheral pain/swelling (BASDAI question 3 result) 0.579 x (natural logarithm of the (hs-CRP [mg/L] + 1)) Back pain, PGADA, duration of morning stiffness, peripheral pain/swelling and fatigue are all assessed on a numerical scale (0 to 10 units).
  The change from Baseline is calculated, a negative value indicating improvement and a positive value worsening. There is a minimum score of 0.636 for the total ASDAS score, but no defined upper score since CRP does not have a set upper limit.
  If one component for the ASDAS-CRP was missing at a given visit, that component was imputed by carrying the last observation forward, and the ASDAS-CRP was calculated accordingly. If the hs-CRP value was below 2 mg/L, then it was imputed as the constant value of 2 mg/L.
Change From Baseline to Week 16 in the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | week 16
  The BASDAI is a validated self-reported instrument, which consists of six 10-unit horizontal Numeric Rating Scales (NRS) to measure severity of fatigue, spinal and peripheral joint pain and swelling, enthesitis, and morning stiffness (both severity and duration, respectively) over the last week. The final BASDAI score ranges from 0 to 10, with lower scores indicating lower disease activity.
  The change from Baseline is calculated, a negative value indicating improvement and a positive value worsening.
  Note: Missing data was imputed using multiple imputation based on the Markov-Chain Monte Carlo method for the intermittent missing data, followed by monotone regression for the monotone missing data assuming missing at random.
Change From Baseline to Week 16 in the Bath Ankylosing Spondylitis Functional Index (BASFI) | week 16
  The BASFI is a validated disease-specific instrument for assessing physical function. The BASFI comprises 10 items relating to the past week. The BASFI is the mean of the 10 scores such that the total score ranges from 0 (Easy) to 10 (Impossible), with lower scores indicating better physical function.
  The change from Baseline is calculated, a negative value indicating improvement and a positive value worsening.
  Note: Missing data was imputed using multiple imputation based on the Markov-Chain Monte Carlo method for the intermittent missing data, followed by monotone regression for the monotone missing data assuming missing at random.
Percentage of Participants With Anti-SCT650C Antibodies | week 52
  A treatment emergent - antidrug antibody (TE-ADA) positive participant is defined as: a) a participant with a >= 4-fold increase over a positive baseline antibody titer; or b) for a negative baseline titer, a participant with an increase from the baseline to a level of >= 1:10. Percentage was calculated based on the number of evaluable participants and was calculated by number of participants with treatment-emergent positive anti-SCT650C antibodies / number of evaluable participants * 100%.
Serum concentrations of SCT650C overtime | week 52
  Serum concentrations of SCT650C overtime

CONTACTS AND LOCATIONS:
Overall Officials: Umut Kalyoncu, Principal Investigator — Hacettepe University Faculty of Medicine, Department of Internal Medicine, Division of Rheumatology
Locations (1):
- Hacettepe University Faculty of Medicine, Ankara, Hacettepe Mh., Turkey (Türkiye)